CLINICAL TRIAL: NCT02863536
Title: A Multicenter, Open Label, Non-comparative, 3 Months Study to Assess the Performance and Safety of the New Medical Device Polybactum® in Reducing the Frequency of Recurrent Bacterial Vaginosis
Brief Title: A Study of the New Medical Device Polybactum®
Acronym: POLARIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Effik Italia S.p.A. (Other)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OPEFF/0116/MD
Record Dates: First submitted 2016-08-01; First posted 2016-08-11 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Bacterial Vaginosis
Keywords: Recurrence of Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Polybactum® (Other): Polybactum® ovules are administered intravaginally on 3 cycles, 1 cycle per month.
  Polybactum is a medical device Class IIa used and marketed for the recurrence of Bacterial Vaginosis.
  Interventions: Device: Polybactum®

INTERVENTIONS:
Device: Polybactum® — 3 cycles treatment one per month.. Duration of one cycle: 1 week; administration for each cycle: 1 ovule at Day 1, 1 ovule at Day 4; 1 ovule at Day 7.In the two following cycles, the same treatment will be repeated immediately after the end of the first and second menstrual bleeding.

SUMMARY:
The POLARIS trial is designed as a multicenter, open label, non-comparative, 3 months, clinical study.

Interventional, non-controlled, multicenter trial with a prospective design on one cohort of patients

DETAILED DESCRIPTION:
To evaluate the efficacy of Polybactum® administered for 3 cycles (one cycle/month) in reducing the rate of recurrence of BV in women cured with vaginal metronidazole and to compare the results of the treatment with the rate of recurrence reported in appropriate selected international literature. Therefore, the Polybactum® early administration should be able to modify the basal individual risk of BV recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Women above 18 years.
* BV diagnosed by Amsel criteria (see Annex 3) in the 6-9 days before study, and cured with metronidazole vaginal formulation (gel for 5 days or ovules for 7 days).
* Diagnosis of RBV (at least 2 episodes of BV in the last 12 months including the BV cured before baseline).
* Non lactating women or lactating non amenorrheic women.
* Read and signed informed consent.

Exclusion Criteria:

* Pregnancy.
* Candidiasis or mixed vaginitis.
* HIV or other immunodeficiency.
* Known allergy to metronidazole or to Polybactum® ingredients.
* Sex workers.
* Menstruation or pre-menopause/menopause.
* Patients concomitantly included in different interventional clinical trials.
* Unwillingness to provide the informed consent to the trial.
* Time between the last day of last menses and baseline visit > 16 days or ≤5 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Amsel criteria laboratory diagnostic | 3 months
  Signs and symptoms of Bacterial Vaginosis assesed also by patients diary (vaginal discharge, burning, erythema, dyspareunia)

SECONDARY OUTCOMES:
Lactobacilli counting | 3 months
  The rate of return to normality of vaginal microflora through Lactobacilli counting

OTHER OUTCOMES:
Patient's diary | 3 months
  Global Assessment of Efficacy by Patient's diary

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Murina, Prof.dr., Principal Investigator — Servizio di Patologia del Tratto Genitale Inferiore U.O. Ostetricia e Ginecologia Ospedale Vittore Buzzi - Universita' degli Studi di Milano Milano (Italy)
Locations (1):
- Opera Contract Research Organization Srl, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwebke JR. Bacterial vaginosis--more questions than answers. Genitourin Med. 1997 Oct;73(5):333-4. doi: 10.1136/sti.73.5.333. No abstract available. PMID 9534738
- [Background] Sobel JD. Antibiotic consideration in bacterial vaginosis. Curr Infect Dis Rep. 2009 Nov;11(6):471-5. doi: 10.1007/s11908-009-0068-5. PMID 19857387
- [Background] Marrazzo JM. Interpreting the epidemiology and natural history of bacterial vaginosis: are we still confused? Anaerobe. 2011 Aug;17(4):186-90. doi: 10.1016/j.anaerobe.2011.03.016. Epub 2011 Apr 16. PMID 21524714
- [Background] Bradshaw CS, Morton AN, Hocking J, Garland SM, Morris MB, Moss LM, Horvath LB, Kuzevska I, Fairley CK. High recurrence rates of bacterial vaginosis over the course of 12 months after oral metronidazole therapy and factors associated with recurrence. J Infect Dis. 2006 Jun 1;193(11):1478-86. doi: 10.1086/503780. Epub 2006 Apr 26. PMID 16652274
- [Background] Donders GG. Definition and classification of abnormal vaginal flora. Best Pract Res Clin Obstet Gynaecol. 2007 Jun;21(3):355-73. doi: 10.1016/j.bpobgyn.2007.01.002. Epub 2007 Apr 16. PMID 17434799
- [Background] Kovachev S, Dobrevski-Vacheva R. [Probiotic monotherapy of bacterial vaginosis: a open, randomized trial]. Akush Ginekol (Sofiia). 2013;52 Suppl 1:36-42. Bulgarian. PMID 24294744
- [Background] Falagas M, Betsi GI, Athanasiou S. Probiotics for the treatment of women with bacterial vaginosis. Clin Microbiol Infect. 2007 Jul;13(7):657-64. doi: 10.1111/j.1469-0691.2007.01688.x. PMID 17633390
- [Background] Vujic G, Jajac Knez A, Despot Stefanovic V, Kuzmic Vrbanovic V. Efficacy of orally applied probiotic capsules for bacterial vaginosis and other vaginal infections: a double-blind, randomized, placebo-controlled study. Eur J Obstet Gynecol Reprod Biol. 2013 May;168(1):75-9. doi: 10.1016/j.ejogrb.2012.12.031. Epub 2013 Feb 7. PMID 23395559
- [Background] Swidsinski A, Mendling W, Loening-Baucke V, Ladhoff A, Swidsinski S, Hale LP, Lochs H. Adherent biofilms in bacterial vaginosis. Obstet Gynecol. 2005 Nov;106(5 Pt 1):1013-23. doi: 10.1097/01.AOG.0000183594.45524.d2. PMID 16260520
- [Background] Senok AC, Verstraelen H, Temmerman M, Botta GA. Probiotics for the treatment of bacterial vaginosis. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD006289. doi: 10.1002/14651858.CD006289.pub2. PMID 19821358
- [Background] Brown P, Brunnhuber K, Chalkidou K, Chalmers I, Clarke M, Fenton M, Forbes C, Glanville J, Hicks NJ, Moody J, Twaddle S, Timimi H, Young P. How to formulate research recommendations. BMJ. 2006 Oct 14;333(7572):804-6. doi: 10.1136/bmj.38987.492014.94. PMID 17038740
- [Background] Pirotta M, Fethers KA, Bradshaw CS. Bacterial vaginosis - More questions than answers. Aust Fam Physician. 2009 Jun;38(6):394-7. PMID 19521581
- [Derived] Murina F, Inghirami P, Biris M, Sirbu D, Barattini DF, Sbrocca F, Ardolino LI, Mangrella M, Casolati E, Rosu S, Crisan CD. Performance and Safety of a New Medical Device (Polybactum) for Reducing the Recurrence Rate of Bacterial Vaginosis: Protocol for a Multicenter, Open-Label, Noncontrolled International Clinical Trial (POLARIS Study). JMIR Res Protoc. 2023 Jul 20;12:e42787. doi: 10.2196/42787. PMID 37471117